CLINICAL TRIAL: NCT03041896
Title: Retrospective Evaluation of the Clinical and Radiographic Performance of Coflex® Interlaminer Technology Versus Decompression With or Without Fusion.
Brief Title: Retrospective Evaluation of Performance of Coflex® Interlaminer Technology Versus Decompression With or Without Fusion
Status: Completed | Type: Observational
Sponsor: Paradigm Spine (Industry)
Collaborators: MCRA (Industry)
Responsible Party: Sponsor
Other Study IDs: CRDC2016
Record Dates: First submitted 2016-10-06; First posted 2017-02-03 (Estimated); Results first posted 2020-05-19 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Spinal Stenosis
MeSH Terms: conditions — Spinal Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Decompression: Standard of care decompression for spinal stenosis, 1 or 2 levels.
  Interventions: Device: coflex® Interlaminar Technology
- Fusion: Standard pedical and rod fixation with standard decompression, 1 or 2 levels.
  Interventions: Device: coflex® Interlaminar Technology
- coflex®: Decompression surgery with the coflex® Interlaminar Technology, 1 or 2 levels.
  Interventions: Device: coflex® Interlaminar Technology
- Hybrid: coflex and fusion at adjacent levels
  Interventions: Device: coflex® Interlaminar Technology

INTERVENTIONS:
Device: coflex® Interlaminar Technology — Interlaminer Technology

SUMMARY:
To evaluate clinical, radiologic and patient-reported outcomes who have been treated 1 or 2 levels with the coflex® Interlaminar Technology or decompression with or without fusion.

DETAILED DESCRIPTION:
The coflex® Interlaminar Technology - manufactured by Paradigm Spine - is intended for use as a permanent implant between the lamina of 1 or 2 lumbar motion segments in the treatment of moderate to severe lumbar spinal stenosis. The device is specifically designed to provide stabilization without fusion in cases of stenosis with or without facet joint hypertrophy, subarticular recess stenosis or foraminal stenosis. It is restricted for use to one or two levels in the region of L1 - L5.

The height of the neuroforamen is maintained and the facet joints will be relieved. By this a further destruction is prevented. Unlike conventional stabilization methods as for example spinal fusion, the function of the segment will be maintained and adjacent structures will be effectively protected.

Possible risks, which could occur after implantation of the coflex® Interlaminar Technology are breakage of the implant, displacement of the implant, pain which is caused by the implant, infections, bleedings and hematoma. The benefit of the study lies in the fact that first-time retrospective data is raised for potential improvement regarding therapy of lumbar back pain with the treatment of the lumbar spinal stenosis, which, in the future, can lead to an improvement of the therapy.

In this study, Paradigm Spine will retrospectively collect clinical and radiographic data for patients treated with the coflex® Interlaminar Technology during normal conditions of use. This data will provide evidence to support publications and marketing.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet the criteria specified in the device labeling including radiographic confirmation of at least moderate lumbar stenosis, which narrows the central spinal canal at one or two contiguous levels from L1-L5 that require surgical decompression.

Exclusion Criteria:

* There are no exclusion criteria's for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients must meet the criteria specified in the device labeling including radiographic confirmation of at least moderate lumbar stenosis, which narrows the central spinal canal at one or two contiguous levels from L1-L5 that require surgical decompression.
Sampling Method: Non-Probability Sample
Enrollment: 5050 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abigail Allen, Study Director — MCRA

IPD SHARING:
Plan to Share IPD: Yes
There are no benefits to the subject as this data is being collected to obtain additional clinical evidence to support publications and marketing.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Decompression | Fusion | Coflex® | Hybrid
Started | 1486 | 1009 | 2299 | 256
Completed | 1486 | 1009 | 2236 | 253
Not Completed | 0 | 0 | 63 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Decompression | Fusion | Coflex® | Hybrid | Total
Number analyzed (Participants) | 1486 | 1009 | 2299 | 256 | 5050
Age, Customized [Mean (Standard Deviation); unit: years]
  Age | 61.9 (15.46) | 65.4 (11.54) | 68.1 (9.96) | 65.8 (10.34) | 65.6 (12.5)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 856 | 402 | 1257 | 137 | 2652
  Female | 629 | 607 | 1040 | 119 | 2395
  Unknown | 1 | 0 | 2 | 0 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 93 | 21 | 40 | 8 | 162
  Not Hispanic or Latino | 564 | 196 | 539 | 25 | 1324
  Unknown or Not Reported | 829 | 792 | 1720 | 223 | 3564
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Black or African American | 80 | 36 | 81 | 14 | 211
  Race: White | 789 | 251 | 1009 | 53 | 2102
  Race: Asian | 5 | 4 | 6 | 0 | 15
  Race: American Indian or Alaska Native | 4 | 1 | 5 | 0 | 10
  Race: Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 1
  Race: Not Specified | 607 | 717 | 1198 | 189 | 2711

OUTCOME MEASURES:

1. Primary Outcome: Overall Duration of Follow-up Care to Evaluate Overall Effectiveness of the Use of the Coflex® Interlaminer Technology
Description: To assess the overall duration of follow-up care to evaluate overall effectiveness of the use of the coflex® Interlaminer Technology verses decompression.
Time Frame: Study Duration Up to 6 months for data collection
Population: The following arms: coflex® and Decompression, were the only arms where this data was collected and compared for this study.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Coflex® | Decompression
Number analyzed (Participants) | 2058 | 1428
days | 201.26 (208.64) | 191.75 (247.23)

2. Primary Outcome: Overall Incidence of Secondary Surgical Interventions Post Surgeries.
Description: To analyze the incidence of secondary surgical interventions to evaluate overall effectiveness of the use of the coflex® Interlaminer Technology vs. decompression.
Time Frame: Study Duration up to 6 months data
Population: The following arms: coflex® , Fusion, and Decompression, were the only arms where this data was collected and compared for this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Decompression | Coflex® | Fusion
Number analyzed (Participants) | 1428 | 2058 | 1009
Participants | 126 | 125 | 99

3. Secondary Outcome: The Secondary Objectives Include Measuring and Comparing Clinical, Radiologic, and Patient Reported Outcomes at Baseline, Interim and/or Final Follow-up Visits.
Description: To assess the impact of demographics and risk factors on clinical, radiologic, and patient reported outcomes, and to assess the operative details and safety outcomes associated with the use of the device.
  The clinical outcomes will be summarized; however, since the collection of these measures is not standard of care, this data will only be collected as available. In addition, data will be used to analyze the association between coflex® Interlaminar Technology use and outcomes with age, race, workers' compensation, smoking status, and gender.
Time Frame: Study Duration Up to 6 months for data collection
Population: The data (clinical, radiologic, and PROs) was not collected from the sites.
Arm/Group | Decompression | Fusion | Coflex® | Hybrid
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Not applicable as safety data were not collected during the study.
Description: No formal analysis of adverse events was performed.
Arm/Group | Decompression | Fusion | Coflex® | Hybrid
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-02): https://cdn.clinicaltrials.gov/large-docs/96/NCT03041896/Prot_SAP_000.pdf